CLINICAL TRIAL: NCT06868849
Title: An Open-label, Multi-center, Phase I Study to Investigate Safety, Tolerability, Pharmacokinetics, and Efficacy of JMT203 in Patients With Cancer Cachexia
Brief Title: A Study of JMT203 in Patients With Cancer Cachexia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMT203-001
Record Dates: First submitted 2025-02-18; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer; Non Small Cell Lung Cancer; Pancreatic Cancer; Cancer Cachexia
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: There is no comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Dose Escalation, Dose Expansion and Cohort Expansion Phase (Experimental): Dose escalation - Five dose levels of JMT203 will be tested in patients with cancer cachexia according to an accelerated titration design combined with a "3+3" dose escalation scheme. If the highest predefined dose group demonstrates good safety and tolerability during dose escalation, further discussion will be held on whether to proceed to a higher dose group or to explore doses between two existing groups.
  Dose expansion - Based on pharmacokinetics (PK), pharmacodynamics (PD), preliminary efficacy, and safety data, 1 to 3 dose levels that are potentially effective will be selected.
  Cohort expansion- There are three cohorts:
  Cohort A: Patients with non-resectable, advanced, recurrent, or metastatic non-small cell lung cancer cachexia.
  Cohort B: Patients with non-resectable, advanced, recurrent, or metastatic pancreatic cancer cachexia.
  Cohort C: Patients with non-resectable, advanced, recurrent, or metastatic colorectal cancer and other types of cachexia.
  Patients with select so
  Interventions: Drug: JMT203 Injection

INTERVENTIONS:
Drug: JMT203 Injection — Drug：JMT203 Injection
  * Anti-GFRAL monoclonal antibody
  * Will be injected subcutaneously once per cycle (3 weeks, on Day 1) for 12 weeks, or will be injected subcutaneously once per cycle (3 weeks, on Day 1).

SUMMARY:
This is an open-label, multicenter Phase I clinical study aimed at evaluating the safety/tolerability, pharmacokinetics, and effectiveness of JMT203 in patients with cancer cachexia.

DETAILED DESCRIPTION:
This is a study of JMT203 in patients with cancer cachexia, comprising two parts: Phase Ia, which involves a dose-escalation and dose-expansion study of JMT203 in patients with cancer cachexia, and Phase Ib, which is a cohort-expansion study of JMT203 in the same patient population. The primary objectives of Phase Ia are to assess the safety/tolerability of JMT203 in patients with cancer cachexia and to determine the maximum tolerated dose (MTD) (if any) and/or the recommended dose for expansion (RDE) of JMT203. In Phase Ib, the primary objectives include evaluating the preliminary efficacy of JMT203 in treating cancer cachexia and determining the recommended Phase 2 dose (RP2D) of JMT203.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Age ≥ 18 years old;
2. Voluntarily participate in the study and sign the informed consent form;
3. Malignant solid tumors confirmed histologically or cytologically, with ongoing or completed anti-tumor treatment, and no significant tumor progression within 28 days prior to the first drug administration:

   * Dose escalation and expansion phase (Phase Ia): The investigator predicts that there will be no need to change the anti-tumor treatment regimen due to disease progression within the first dosing cycle (21 days) of this study;
   * Cohort expansion study phase (Phase Ib): Cohorts A/B/C will enroll patients with non-small cell lung cancer, pancreatic cancer, and colorectal cancer, respectively;
4. Diagnosed with cancer cachexia according to the criteria of the 2011 International Consensus on Cancer Cachexia: Definition and Classification, combined with characteristics of the Chinese population, i.e., presenting with one of the following within 6 months (previous weight data must be supported by written documentation approved by the sponsor): involuntary weight loss >5%, or weight loss >2% when Body Mass Index （BMI） <18.5 kg/m²;
5. Serum Growth Differentiation Factor 15 （GDF-15） levels ≥1300 pg/ml within 28 days prior to the first study drug administration (applicable to the cohort expansion phase only);
6. Adequate organ function, meeting relevant laboratory test standards:

   Item Laboratory Test Value Blood Absolute Neutrophil Count ≥1.0×10^9/L Platelet Count ≥75×10^9/L Hemoglobin ≥80 g/L Kidney Serum Creatinine ≤1.5×ULN (if >1.5×ULN, creatinine clearance calculated by the Cockcroft formula must≥30 ml/min) Liver Total Bilirubin ≤1.5×ULN (For patients with liver metastasis, liver cancer, or bile duct obstruction: may be relaxed to ≤3×ULN) AST and ALT ≤3×ULN or ≤5×ULN for patients with liver metastasis Coagulation APTT ≤1.5×ULN INR ≤1.5×ULN Note: ULN = Upper Limit of Normal; if laboratory tests do not meet the criteria, the investigator will determine eligibility based on the patient's overall condition.
7. 7. Eastern Cooperative Oncology Group Performance Status （ECOG PS）score: ≤2;
8. Estimated survival ≥4 months;
9. Fertile eligible patients must use adequate contraceptive measures from the time of signing the informed consent form until 6 months after the last drug administration; female patients of childbearing age must have a negative serum pregnancy test within 7 days before the first drug administration.

Exclusion Criteria:

1. Presence of reversible causes leading to decreased food intake;
2. Patients with dysphagia or poor food digestion and absorption, including gastrointestinal obstruction, active inflammatory bowel disease, or short bowel syndrome;
3. Patients with cachexia caused by clearly identified other causes, such as severe chronic obstructive pulmonary disease, uncontrolled thyroid disease, vital organ failure, or Acquired Immune Deficiency Syndrome （AIDS）;
4. Patients receiving tube feeding or parenteral nutrition therapy during the screening period;
5. Patients who have taken any prescription medications for appetite enhancement or improve weight loss within 28 days or 5 half-lives (whichever is shorter) before the first study drug administration, including but not limited to anamorelin, medroxyprogesterone acetate, dronabinol, medical marijuana, etc.;
6. Initiation of systemic glucocorticoids (prednisone >10 mg/day or equivalent doses of other similar drugs) or other immunosuppressive therapies within 28 days before the first study drug administration, excluding pretreatment for antitumor therapy;
7. Patients with a BMI exceeding 30 kg/m²;
8. Patients who have undergone major surgery within 4 weeks before the first study drug administration and have not recovered, or are expected to undergo major surgery during the study;
9. Patients who have received other clinical study medications within 4 weeks or 5 half-lives (whichever is shorter) before the first study drug administration;
10. Patients with severe infections requiring intravenous antibiotics, antivirals, or antifungals during the screening period;
11. Patients with difficult-to-control moderate to large amounts of serous cavity effusion, such as pericardial effusion or pleural/abdominal/pelvic effusion, within 14 days before the first study drug administration;
12. Patients with a second primary active malignancy within 2 years before the first study drug administration, excluding locally curable tumors that have undergone radical treatment (e.g., resected basal cell or squamous cell skin cancer, superficial bladder cancer, breast carcinoma in situ);
13. Patients with active central nervous system metastases (brain metastases, carcinomatous meningitis, and spinal cord metastases), except for those with controlled lesions confirmed by imaging studies within 28 days before the first use of the investigational product;
14. History of severe cardiovascular disease, including but not limited to:

    1. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, second- or third-degree atrioventricular block, etc.;
    2. Occurrence of acute coronary syndrome, congestive heart failure, stroke, or other cardiovascular events of grade 3 or higher within 6 months before the first study drug administration;
    3. New York Heart Association functional class ≥III or left ventricular ejection fraction (LVEF) <50%;
15. Patients with severe immune deficiency or a history of organ transplantation;
16. Patients with recent (within the past year) or current depression or suicidal ideation/tendencies;
17. Known allergy to JMT203 or its components;
18. History of severe allergic reactions or uncontrollable allergic asthma;
19. Patients deemed unsuitable for participation in this clinical study by the investigator for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs). | Up to 90 days after the last dose of JMT203
Phase Ia: Incidence of dose-limiting toxicity (DLT) events | Up to 21 days after the first dose of JMT203
Phase Ia: MTD (if applicable). | Up to 90 days post last dose
Phase Ia: RDE. | Up to 90 days post last dose
Phase Ib: Average change in body weight from baseline at each assessment timepoint within 12 weeks. | Within 12 weeks from baseline

SECONDARY OUTCOMES:
Phase Ia: Area under the curve from time "0" to the time of the last measurable concentration (AUC0-t) of JMT203 | Up to 90 days after the last dose of JMT203
Phase Ia: Maximum measured plasma concentration (Cmax) of JMT203 | Up to 90 days after the last dose of JMT203
Phase Ia: Time when Cmax occurred (Tmax) of JMT203 | Up to 90 days after the last dose of JMT203
Phase Ia: The PD indicators include β-hydroxybutyric acid. | Up to 12 weeks
Phase Ia: Incidence of anti-drug antibodies (ADA). | Up to 90 days after the last dose of JMT203
Phase Ia: Average change in body weight from baseline at each assessment timepoint within 12 weeks | Within 12 weeks from baseline
Phase Ib: Average change in the skeletal muscle index (SMI) of the third lumbar vertebra, measured by computed tomography (CT), from baseline to 12 weeks. | Within 12 weeks from baseline
Phase Ib: Average change in the severity of anorexia (based on the Functional Assessment of Anorexia/Cachexia Therapy - Anorexia/Cachexia Subscale [FAACT-A/CS]) from baseline to each assessment timepoint. | Within 12 weeks from baselineUp until the end of the treatment
Phase Ib: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs). | Up to 90 days after the last dose of JMT203
Phase Ib: Blood concentration of JMT203; | Up to 90 days after the last dose of JMT203
Phase Ib: PD indicators include β-hydroxybutyric acid. | Up to 24 weeks
Phase Ib: Incidence of ADA. | Up to 90 days after the last dose of JMT203
Phase Ib: overall survival (OS). | Approximately up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sir run run shaw Hospital, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No